CLINICAL TRIAL: NCT02813551
Title: Torsemide for the Prevention of Persistent Postpartum Hypertension in Preeclamptic Women: A Randomized, Placebo-Control Trial
Brief Title: ToRsemide for pOstpartum HYpertension
Acronym: TROPHY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Oscar Andres Viteri Molina, Maternal-Fetal Medicine Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC-MS-16-0198
Record Dates: First submitted 2016-06-19; First posted 2016-06-27 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Preeclampsia
Keywords: Preeclampsia, puerperium
MeSH Terms: conditions — Pre-Eclampsia | interventions — Torsemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Torsemide (Experimental): Torsemide 20 mg daily for 5 days
  Interventions: Drug: Torsemide
- Placebo (Placebo Comparator): Placebo 20 mg daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Torsemide
  Other Names: Demadex, torasemide
  Arms: Torsemide
Drug: Placebo
  Arms: Placebo

SUMMARY:
Currently there is no intervention to prevent persistent postpartum hypertension in preeclamptic women. Physiologically, the use of a pharmacokinetically predictable loop-diuretic is a reasonable intervention to increase elimination of extra fluid accumulated secondary to preeclampsia.The purpose of this study is to assess if Torsemide reduces the incidence of persistent postpartum hypertension in preeclamptic women.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women at ≥ 18 years of age
* Antepartum/intrapartum or within 24 hours postpartum diagnosis of either:
* Preeclampsia
* Preeclampsia with severe features
* Preeclampsia superimposed to chronic hypertension

Exclusion Criteria:

* Chronic hypertension without superimposed preeclampsia
* Gestational hypertension
* Urine output < 30 cc/h at time of randomization
* Heart failure or pulmonary edema
* Hypersensitivity to Torsemide or sulfonylureas
* Hypokalemia (serum potassium < 3 mEq/L)
* Preexisting diuretic use within 24 hours prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07-28 (Actual); Study Completion 2017-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Viteri OA, Alrais MA, Pedroza C, Hutchinson M, Chauhan SP, Blackwell SC, Sibai BM. Torsemide for Prevention of Persistent Postpartum Hypertension in Women With Preeclampsia: A Randomized Controlled Trial. Obstet Gynecol. 2018 Nov;132(5):1185-1191. doi: 10.1097/AOG.0000000000002941. PMID 30303905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Torsemide | Placebo
Started | 59 | 59
Completed | 58 | 57
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Torsemide | Placebo | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (6.1) | 28.2 (6.8) | 27.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 13 | 29
  Not Hispanic or Latino | 43 | 46 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 33 | 35 | 68
  Race: Caucasian | 9 | 11 | 20
  Race: Hispanic | 16 | 13 | 29
  Race: Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 59 | 118
Body Mass Index (BMI) at delivery [Mean (Standard Deviation); unit: kg/m^2] | 38.3 (10.4) | 37.0 (9.9) | 37.7 (10.2)
Married [Count of Participants; unit: Participants] | 21 | 20 | 41
Nulliparous [Count of Participants; unit: Participants] | 38 | 31 | 69
Smoker [Count of Participants; unit: Participants] | 1 | 5 | 6
Use of illicit drugs [Count of Participants; unit: Participants] | 6 | 5 | 11
Use of Cocaine [Count of Participants; unit: Participants] | 1 | 0 | 1
Prenatal care [Count of Participants; unit: Participants] | 59 | 55 | 114
Form of Payment [Count of Participants; unit: Participants]
  Government/Subsidized Insurance | 46 | 44 | 90
  Private Insurance | 12 | 14 | 26
  None/Self Paid | 1 | 1 | 2
Pregestational Diabetes [Count of Participants; unit: Participants] | 7 | 6 | 13
Gestational Diabetes [Count of Participants; unit: Participants] | 5 | 5 | 10
Chronic Hypertension [Count of Participants; unit: Participants] | 15 | 15 | 30
Asthma [Count of Participants; unit: Participants] | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Persistent Postpartum Hypertension Defined as Systolic Blood Pressure ≥ 150 and/or Diastolic Blood Pressure ≥ 100 mmHg
Description: Persistent postpartum hypertension was defined as sustained systolic blood pressure ≥ 150 or diastolic blood pressure ≥ 100 mmHg by postpartum day 5 or at hospital discharge, whichever occurred first.
Time Frame: 0-5 days after delivery
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 26 | 34
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.53 to 1.10]

2. Secondary Outcome: Number of Participants With Severe Postpartum Hypertension Requiring Acute Antihypertensives (Systolic Blood Pressure ≥160 and/or Diastolic Blood Pressure ≥ 110 mmHg)
Time Frame: 0-6 weeks after delivery
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 7 | 6
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.4 to 3.3]

3. Secondary Outcome: Number of Participants Requiring Postpartum Readmission
Time Frame: 0-6 weeks after delivery
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 3 | 1
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 3.0, 95% CI 2-sided [0.3 to 28]

4. Secondary Outcome: Length of Hospital Stay After Delivery
Time Frame: 0-5 days after delivery
Population: Intention-to-treat
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
hours | 68 [52 to 94] | 54 [47 to 77]
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.1, 95% CI 2-sided [1.0 to 1.3]

5. Secondary Outcome: Weight Change
Time Frame: at the time of randomization (within 24 hours of delivery); at discharge (about 1-5 days after delivery)
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
pounds | 3.01 (3.85) | 2.08 (2.69)

6. Secondary Outcome: Change in Lower Extremity Edema
Description: Lower extremity edema was assessed by measuring right ankle circumference at 5 centimeters above the medial malleolus.
Time Frame: at the time of randomization (within 24 hours of delivery); at discharge (about 1-5 days after delivery)
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
millimeters | -1.29 (12.08) | -2.9 (14.08)

7. Secondary Outcome: Number of Participants With Persistent Postpartum Hypertension (Systolic Blood Pressure ≥140 and/or Diastolic Blood Pressure ≥ 90 mmHg)
Time Frame: 7-10 days after delivery
Population: 38 (42%) women in the torsemide group and 31 (53%) women in the placebo missed their outpatient clinic visit at 7-10 days after delivery, resulting in only 21 in the torsemide group and 28 in the placebo group being analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 21 | 28
Participants | 9 | 11
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.1, 95% CI 2-sided [1.0 to 1.2]

8. Secondary Outcome: Number of Participants With Persistent Postpartum Hypertension (Systolic Blood Pressure ≥140 and/or Diastolic Blood Pressure ≥ 90 mmHg)
Time Frame: 6 weeks after delivery
Population: 36 women in the torsemide group and 28 women in the placebo group did not show to their clinic appointment 6 weeks after delivery, resulting in 23 in the torsemide group and 31 in the placebo group being analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 23 | 31
Participants | 8 | 11
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.5 to 1.9]

9. Secondary Outcome: Number of Participants With Side Effects of Therapy - Hypokalemia (Low Blood Potassium Levels)
Time Frame: 0-5 days after delivery
Population: Blood potassium levels were only collected for 22 in the torsemide group and 31 in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 22 | 31
Participants | 1 | 4
Statistical Analysis 1: Comparison: Torsemide vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.4, 95% CI 2-sided [0.1 to 2.9]

10. Secondary Outcome: Number of Participants With Side Effects of Therapy - Decreased Breast Milk
Time Frame: 0-5 days after delivery
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 1 | 0

11. Secondary Outcome: Number of Participants With Severe Composite Maternal Morbidity
Description: Severe composite maternal morbidity is defined as having any of the following: ICU admission, HELLP syndrome, eclampsia, stroke, renal failure, pulmonary edema, cardiomyopathy, or maternal death.
Time Frame: 0-6 weeks after delivery
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 0 | 0

12. Other Pre Specified Outcome: Torsemide Concentrations in Breast Milk
Description: Ancillary study
Time Frame: 0-5 days after delivery
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Electrolyte Profile in Maternal Serum
Description: Concentrations of: Sodium, Potassium, Calcium
Time Frame: 0-5 days after delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Only related adverse events were recorded. Blood potassium levels were only collected for 22 in the torsemide group and 31 in the placebo group, thus only 22 in the torsemide group and 31 in the placebo group are indicated as at risk for hypokalemia.
Arm/Group | Torsemide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 2/59 | 4/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Torsemide (N=59) | Placebo (N=59)
Hypokalemia (low blood potassium levels) (General disorders) | 1/22 (1) | 4/31 (4)
Decreased breast milk (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Median hospital stay <3 days, but sample size powered to detect differences in up to 5 days. High rate of clinic no-shows. Not powered to detect differences in secondary outcomes. Edema measurements done with stocking, which may affect reliability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02813551/Prot_SAP_000.pdf